CLINICAL TRIAL: NCT00136526
Title: Docetaxel and Diethylstilbestrol in the Treatment of Androgen Independent Prostate Cancer: A Phase II Study
Brief Title: Docetaxel and Diethylstilbestrol in the Treatment of Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-4599-V; FHCRC-UW-02-4599-V
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Hormone refractory prostate cancer; Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Diethylstilbestrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel and Diethylstilbestrol (DES) — Subjects receive docetaxel 36 Mg/m2weekly for ten cycles (3 weeks out of every 4) and DES 1 mg daily for 40 weeks or until there is evidence of disease progression, whichever occurs first.

SUMMARY:
This study is for men who have prostate cancer that has spread outside of the prostate gland and is no longer responding to hormone removal therapy. This study is designed to determine if a new drug combination will help to control the cancer. The medicines being used, docetaxel and diethylstilbestrol (DES), have been given to patients with prostate cancer and each drug has demonstrated activity in prostate cancer, either used alone or in other combinations. The objective of this study is to determine the effect of this drug combination on the prostate cancer and its response to disease progression.

DETAILED DESCRIPTION:
This is a single arm phase II trial of docetaxel and diethylstilbestrol for patients with symptomatic stage D3 androgen independent prostate cancer. Patients will receive docetaxel weekly for 10 cycles (each cycle consists of treatment for 3 weeks out of every 4) and DES daily for 40 weeks or until there is evidence of disease progression, whichever occurs first. Patients will be followed to determine PSA and objective response. Additional endpoints include time to progression, disease specific survival and overall survival. Disease progression will be defined as 2 consecutive increases in PSA and/or tumor growth as evidenced by examination or radiologic evaluation. Other secondary objectives will be to determine the toxicity, and impact on quality of life of this regimen.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria are eligible for the trial:

* Men 18 years of age or older with a histologically confirmed diagnosis of adenocarcinoma of the prostate consistent with stage D3.
* Prior therapy with medical or surgical castration and evidence of castrate levels of testosterone
* Discontinuation of nonsteroidal antiandrogens more than 6 weeks prior to evaluation for progression. It is not a requirement that nonsteroidal antiandrogen therapy be used prior to enrollment.
* Androgen independent disease as defined by one of the following after androgen ablation and withdrawal from nonsteroidal antiandrogen if initiated (> 6 weeks after discontinuation):

  * PSA must be greater than 5 ng/ml and increasing as demonstrated by two consecutive increasing PSA levels over 5 ng/ml. Each PSA measurement must be taken at least one week apart.
  * Increase in measurable disease within one month of enrollment
  * Worsening of bone scan abnormalities within two months of enrollment and greater than four months since initiation of luteinizing hormone-releasing hormone (LHRH) agonist.
* Performance status < 3 by the Eastern Cooperative Oncology Group (ECOG) scale.
* Patients must be informed of the investigational nature of the study and sign an informed consent form.
* Life expectancy must be >= 3 months.
* Laboratory values must be as follows:

  * White blood cell count: >= 3,000/mm3
  * Absolute granulocyte count: >= 1,500/mm3
  * Platelets: >= 100,000/mm3
  * Hemoglobin: >= 8g/dL
  * Serum creatinine: <= 1.5 x upper limit of normal (ULN)
  * AST: <= 2 x ULN
  * ALT: <= 2 x ULN
  * Serum calcium: <= ULN
  * Total bilirubin: <= 1.5 x ULN
* Patient must be willing to consent to using effective contraception while on treatment and for three months after completion of therapy.

Exclusion Criteria:

Patients meeting any of the following criteria will not be eligible for the trial:

* Patients who have received PC-SPES, DES, mitoxantrone or docetaxel therapy.
* Patients who have received prior chemotherapy of any type or are receiving any other investigational therapy.
* Patients with evidence of recent deep venous thrombosis, pulmonary emboli, unstable angina or clinical congestive heart failure.
* Patients with a prior history of myocardial infarction, pulmonary embolism, cerebral vascular accident (CVA) or atrial fibrillation.
* Patients with evidence of active angina as evidenced by chest pain responsive to sublingual nitroglycerin or other anginal equivalent.
* Patients with known evidence of brain metastases or carcinomatous meningitis.
* Patients with a history of other cancers except curatively-treated non-melanomatous skin cancer. Other cured tumors may be entered after discussion with and approval of the study chair.
* Patients with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
* Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 must be excluded.
* Histologic evidence of small cell carcinoma of the prostate.
* Patients with current peripheral neuropathy of any etiology that is greater than Grade I.
* Patients with contraindications to anti-coagulation.

Ages: 21 Years to 83 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-12; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Monthly PSA levels and scans every 3 months while on therapy | Over 10 months

SECONDARY OUTCOMES:
To evaluate the time to progression of disease | Follow-up until progression
To determine the risk of cardiovascular complications associated with DES plus aspirin and warfarin 2 mg daily | Over 10 months while on therapy
To measure this regimen's toxicity and impact on quality of life measures | Over 10 months while on therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Montgomery, MD, Principal Investigator — University of Washington